CLINICAL TRIAL: NCT04107584
Title: Prognostic Value of Plasma Biomarkers Among Patients With Hypertension
Acronym: BIOMS-HTN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: HTN2019
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertension is the most important risk factor for cardiovascular and cerebrovascular diseases，and also a substantial public health problem. The purpose of the study is to investigate the association between plasma biomarkers and adverse outcomes in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* In accordance with the diagnosis of hypertension (BP≥140/90mmHg)

Exclusion Criteria:

* The exclusion Criteria for the study program were as follows:

Pregnancy, history of heart failure or left ventricular ejection fraction less than 40%, myocardial infarction within one month, percutaneous transluminal coronary angioplasty or coronary artery bypass grafting, cerebrovascular disease, severe liver disease, severe chronic renal failure (eGFR less than 30 mL/min/1.73 m2) in the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Primary mortality of hypertension | Through study completion, an average of 2 years
  The incidence rate of primary mortality of hypertension

SECONDARY OUTCOMES:
Secondary outcomes of heart | Through study completion, an average of 2 years
  The incidence rate of left ventricular hypertrophy, myocardial infarction, congestive heart failure, and arrhythmia
Secondary outcomes of brain | Through study completion, an average of 2 years
  The incidence rate of stroke (include cerebral hemorrhage and cerebral ischemia
Secondary outcomes of kidney | Through study completion, an average of 2 years
  The incidence rate of hypertensive renal injure and end-stage renal disease
Secondary outcomes of eyes | Through study completion, an average of 2 years
  The incidence rate of hypertensive eye injure

CONTACTS AND LOCATIONS:
Overall Officials: Jie Du, PhD, Study Director — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided